CLINICAL TRIAL: NCT06352372
Title: Safety and Efficacy of Transcranial Photobiomodulation (tPBM) for Individuals With Autism Spectrum Disorder and Epileptiform Activity
Brief Title: Safety and Efficacy of tPBM for Epileptiform Activity in Autism
Acronym: tPBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Frye (Other)
Responsible Party: Sponsor-Investigator, Richard Frye, Principal Investigator and Sponsor, Rossignol Medical Center
Organization: Rossignol Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tPBM Study
Record Dates: First submitted 2024-03-22; First posted 2024-04-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; EEG With Periodic Abnormalities; Epilepsy; Neurodevelopmental Disorders; Neurological Disorder
Keywords: Autism; Epilepsy; Neurological Disorders; Neurodevelopmental disorders; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Epilepsy; Neurodevelopmental Disorders; Nervous System Diseases; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This is a prospective, open label study comparing 15 individuals with active seizures and 15 individuals with EEG abnormalities before and after treatment with, near infra-red (NIR) light - transcranial Photobiomodulation (tPBM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) - to the brain of autistic child (Experimental): This is a prospective, open level study comparing 15 individuals with active seizures and 15 individuals with EEG abnormalities before and after, near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) will be the active arm and the second arm will receive a placebo (no intervention).
  Interventions: Device: noninvasively delivered near infra-red (NIR) light - transcranial Photobiomodulation (tPBM)

INTERVENTIONS:
Device: noninvasively delivered near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) — The proposed intervention will be noninvasively delivered near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) - to the brains of autistic children. The NIR light is delivered to specific brain areas by Cognilum, a wearable device developed by Jelikalite. The expected outcome is improved focus, improved eye contact, improved speech, improved behavior, and gains in functional skills.

SUMMARY:
For this study, the proposed intervention will be noninvasively delivered near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) - to the brains of autistic children. This will occur, twice a week, for 10 weeks. The NIR light is delivered to specific brain areas by Cognilum, a wearable device developed by Jelikalite. The expected outcome is improved focus, improved eye contact, improved speech, improved behavior, and gains in functional skills. Cognilum may impact the clinical practice of treating autism. At the beginning, at five weeks, and at the end of study, the clinician will complete the CARS-2, SRS, CGI, and a caregiver interview; additionally, questionnaires will be administered to caregivers during one of the 1-hour weekly treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (diagnosed as Autistic Disorder on the ADOS-2 or the ADI-R).
* Between 4 and 12 years of age, at baseline.
* Autism severity of moderate or higher (≥4) under the 7-item clinical global impression-severity scale. Moderate level of autism severity (4) is defined by the diagnosis of ASD with language impairment.
* Ability to maintain all ongoing complementary, dietary, traditional, and behavioral treatments constant for the study period.
* Unchanged complementary, dietary, traditional, and behavioral treatments for two months prior to study entry
* Ability to tolerate procedures, as determined at the discretion of the investigator.
* At least one 24hr EEG with data in EDF format that is accessible to investigators.

Exclusion Criteria:

* Significant self-abusive or violent behavior or evidence of suicidal ideation, plan or behavior
* Severely affected children as defined by CGI-Severity Standard Score = 7 (Extremely Ill)
* Severe prematurity (<34 weeks gestation) as determined by medical history
* Current uncontrolled gastroesophageal reflux disease since GERD can cause movements that appear like seizures
* Genetic syndromes
* Congenital brain malformations
* Any medical condition that the PI determines could jeopardize the safety of the study subject or compromise the integrity of the data.
* Failure to thrive or Body Mass Index < 5%ile or <5%ile for weight (male <11.2kg; female <10.8kg by CDC 2000 growth charts) at the time of the study.
* Concurrent treatment with drug that would significantly interact with treatment.

  * • Stimulants
  * • Anti-Psychotics
  * • Antihistamines
* Excessive Hair that the caregivers are unwilling or unable to shave or braid.
* Inability to tolerate the required dosage of tPBM treatment due to sensory issues.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scores (CARS) | Baseline, Week 11 and Week 15 (One Month Follow-Up)
  The CARS is a measure of autism severity completed by a clinician. Lower Score is Better. Scores range from 15 to 60.

SECONDARY OUTCOMES:
EEG Delta Power | Before Treatment and EEG following treatment (within 6 months)
  Delta power is a measures of the amount of brain activity in the delta frequency as measured by overnight EEG

OTHER OUTCOMES:
Seizure frequency and severity | Baseline, Week 11 and Week 15 (One Month Follow-Up)
  Seizure log will record the seizure severity and frequency
Social Responsiveness Scale (SRS) | Baseline, Week 11 and Week 15 (One Month Follow-Up)
  The SRS is a caregiver report of autism symptoms Lower Score is Better, Scores range from 30 to 90 (T-scores)
Clinical Global Impression Scale (CGI) | Baseline, Week 11 and Week 15 (One Month Follow-Up)
  The CGI measures the overall disease severity and change. It is completed by a clinician. Scores range from 1 to 7. Lower score is better
NIH Toolbox | Baseline, Week 11 and Week 15 (One Month Follow-Up)
  The NIH ToolBox is a set of short assessments for neurodevelopmental assessments. Direction of score depends on individual subtest.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, M.D., Ph.D, Principal Investigator — Rossignol Medical Center, Phoenix AZ
Locations (1):
- Rossignol Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett DW, Gonzalez-Lima F. Transcranial infrared laser stimulation produces beneficial cognitive and emotional effects in humans. Neuroscience. 2013 Jan 29;230:13-23. doi: 10.1016/j.neuroscience.2012.11.016. Epub 2012 Nov 27. PMID 23200785
- [Background] Blanco NJ, Maddox WT, Gonzalez-Lima F. Improving executive function using transcranial infrared laser stimulation. J Neuropsychol. 2017 Mar;11(1):14-25. doi: 10.1111/jnp.12074. Epub 2015 May 28. PMID 26017772
- [Background] Cassano P, Petrie SR, Mischoulon D, Cusin C, Katnani H, Yeung A, De Taboada L, Archibald A, Bui E, Baer L, Chang T, Chen J, Pedrelli P, Fisher L, Farabaugh A, Hamblin MR, Alpert JE, Fava M, Iosifescu DV. Transcranial Photobiomodulation for the Treatment of Major Depressive Disorder. The ELATED-2 Pilot Trial. Photomed Laser Surg. 2018 Dec;36(12):634-646. doi: 10.1089/pho.2018.4490. Epub 2018 Oct 20. PMID 30346890
- [Background] Darlot F, Moro C, El Massri N, Chabrol C, Johnstone DM, Reinhart F, Agay D, Torres N, Bekha D, Auboiroux V, Costecalde T, Peoples CL, Anastascio HD, Shaw VE, Stone J, Mitrofanis J, Benabid AL. Near-infrared light is neuroprotective in a monkey model of Parkinson disease. Ann Neurol. 2016 Jan;79(1):59-75. doi: 10.1002/ana.24542. Epub 2015 Dec 12. PMID 26456231
- [Background] Desmet KD, Paz DA, Corry JJ, Eells JT, Wong-Riley MT, Henry MM, Buchmann EV, Connelly MP, Dovi JV, Liang HL, Henshel DS, Yeager RL, Millsap DS, Lim J, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Clinical and experimental applications of NIR-LED photobiomodulation. Photomed Laser Surg. 2006 Apr;24(2):121-8. doi: 10.1089/pho.2006.24.121. PMID 16706690
- [Background] De Taboada L, Yu J, El-Amouri S, Gattoni-Celli S, Richieri S, McCarthy T, Streeter J, Kindy MS. Transcranial laser therapy attenuates amyloid-beta peptide neuropathology in amyloid-beta protein precursor transgenic mice. J Alzheimers Dis. 2011;23(3):521-35. doi: 10.3233/JAD-2010-100894. PMID 21116053
- [Background] Dmochowski GM, Shereen AD, Berisha D, Dmochowski JP. Near-Infrared Light Increases Functional Connectivity with a Non-thermal Mechanism. Cereb Cortex Commun. 2020 Mar 19;1(1):tgaa004. doi: 10.1093/texcom/tgaa004. eCollection 2020. PMID 34296085
- [Background] Giulivi C, Zhang YF, Omanska-Klusek A, Ross-Inta C, Wong S, Hertz-Picciotto I, Tassone F, Pessah IN. Mitochondrial dysfunction in autism. JAMA. 2010 Dec 1;304(21):2389-96. doi: 10.1001/jama.2010.1706. PMID 21119085
- [Background] Hipskind SG, Grover FL Jr, Fort TR, Helffenstein D, Burke TJ, Quint SA, Bussiere G, Stone M, Hurtado T. Pulsed Transcranial Red/Near-Infrared Light Therapy Using Light-Emitting Diodes Improves Cerebral Blood Flow and Cognitive Function in Veterans with Chronic Traumatic Brain Injury: A Case Series. Photomed Laser Surg. 2018 Nov 28. doi: 10.1089/pho.2018.4489. Online ahead of print. PMID 30418082
- [Background] Karu TI, Pyatibrat LV, Afanasyeva NI. Cellular effects of low power laser therapy can be mediated by nitric oxide. Lasers Surg Med. 2005 Apr;36(4):307-14. doi: 10.1002/lsm.20148. PMID 15739174
- [Background] Lampl Y, Zivin JA, Fisher M, Lew R, Welin L, Dahlof B, Borenstein P, Andersson B, Perez J, Caparo C, Ilic S, Oron U. Infrared laser therapy for ischemic stroke: a new treatment strategy: results of the NeuroThera Effectiveness and Safety Trial-1 (NEST-1). Stroke. 2007 Jun;38(6):1843-9. doi: 10.1161/STROKEAHA.106.478230. Epub 2007 Apr 26. PMID 17463313
- [Background] Leisman G, Machado C, Machado Y, Chinchilla-Acosta M. Effects of Low-Level Laser Therapy in Autism Spectrum Disorder. Adv Exp Med Biol. 2018;1116:111-130. doi: 10.1007/5584_2018_234. PMID 29956199
- [Background] Maiello M, Losiewicz OM, Bui E, Spera V, Hamblin MR, Marques L, Cassano P. Transcranial Photobiomodulation with Near-Infrared Light for Generalized Anxiety Disorder: A Pilot Study. Photobiomodul Photomed Laser Surg. 2019 Oct;37(10):644-650. doi: 10.1089/photob.2019.4677. PMID 31647775
- [Background] Naeser MA, Zafonte R, Krengel MH, Martin PI, Frazier J, Hamblin MR, Knight JA, Meehan WP 3rd, Baker EH. Significant improvements in cognitive performance post-transcranial, red/near-infrared light-emitting diode treatments in chronic, mild traumatic brain injury: open-protocol study. J Neurotrauma. 2014 Jun 1;31(11):1008-17. doi: 10.1089/neu.2013.3244. Epub 2014 May 8. PMID 24568233
- [Background] Naeser MA, Martin PI, Ho MD, Krengel MH, Bogdanova Y, Knight JA, Yee MK, Zafonte R, Frazier J, Hamblin MR, Koo BB. Transcranial, Red/Near-Infrared Light-Emitting Diode Therapy to Improve Cognition in Chronic Traumatic Brain Injury. Photomed Laser Surg. 2016 Dec;34(12):610-626. doi: 10.1089/pho.2015.4037. PMID 28001756
- [Background] Naeser MA, Ho MD, Martin PI, Hamblin MR, Koo BB. Increased Functional Connectivity Within Intrinsic Neural Networks in Chronic Stroke Following Treatment with Red/Near-Infrared Transcranial Photobiomodulation: Case Series with Improved Naming in Aphasia. Photobiomodul Photomed Laser Surg. 2020 Feb;38(2):115-131. doi: 10.1089/photob.2019.4630. Epub 2019 Oct 17. PMID 31621498
- [Background] Ortiz-Mantilla S, Cantiani C, Shafer VL, Benasich AA. Minimally-verbal children with autism show deficits in theta and gamma oscillations during processing of semantically-related visual information. Sci Rep. 2019 Mar 25;9(1):5072. doi: 10.1038/s41598-019-41511-8. PMID 30911038
- [Background] Purushothuman S, Johnstone DM, Nandasena C, Mitrofanis J, Stone J. Photobiomodulation with near infrared light mitigates Alzheimer's disease-related pathology in cerebral cortex - evidence from two transgenic mouse models. Alzheimers Res Ther. 2014 Jan 3;6(1):2. doi: 10.1186/alzrt232. eCollection 2014. PMID 24387311
- [Background] Reinhart F, Massri NE, Torres N, Chabrol C, Molet J, Johnstone DM, Stone J, Benabid AL, Mitrofanis J, Moro C. The behavioural and neuroprotective outcomes when 670nm and 810nm near infrared light are applied together in MPTP-treated mice. Neurosci Res. 2017 Apr;117:42-47. doi: 10.1016/j.neures.2016.11.006. Epub 2016 Nov 18. PMID 27871905
- [Background] Salgado AS, Zangaro RA, Parreira RB, Kerppers II. The effects of transcranial LED therapy (TCLT) on cerebral blood flow in the elderly women. Lasers Med Sci. 2015 Jan;30(1):339-46. doi: 10.1007/s10103-014-1669-2. Epub 2014 Oct 3. PMID 25277249
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Wan S, Anderson RR, Parrish JA. Analytical modeling for the optical properties of the skin with in vitro and in vivo applications. Photochem Photobiol. 1981 Oct;34(4):493-9. doi: 10.1111/j.1751-1097.1981.tb09391.x. PMID 7312955
- [Background] Wong-Riley MT, Liang HL, Eells JT, Chance B, Henry MM, Buchmann E, Kane M, Whelan HT. Photobiomodulation directly benefits primary neurons functionally inactivated by toxins: role of cytochrome c oxidase. J Biol Chem. 2005 Feb 11;280(6):4761-71. doi: 10.1074/jbc.M409650200. Epub 2004 Nov 22. PMID 15557336
- [Background] Zivin JA, Sehra R, Shoshoo A, Albers GW, Bornstein NM, Dahlof B, Kasner SE, Howard G, Shuaib A, Streeter J, Richieri SP, Hacke W; NEST-3 investigators. NeuroThera(R) Efficacy and Safety Trial-3 (NEST-3): a double-blind, randomized, sham-controlled, parallel group, multicenter, pivotal study to assess the safety and efficacy of transcranial laser therapy with the NeuroThera(R) Laser System for the treatment of acute ischemic stroke within 24 h of stroke onset. Int J Stroke. 2014 Oct;9(7):950-5. doi: 10.1111/j.1747-4949.2012.00896.x. Epub 2012 Sep 27. PMID 23013107
- [Background] Zomorrodi R, Loheswaran G, Pushparaj A, Lim L. Pulsed Near Infrared Transcranial and Intranasal Photobiomodulation Significantly Modulates Neural Oscillations: a pilot exploratory study. Sci Rep. 2019 Apr 19;9(1):6309. doi: 10.1038/s41598-019-42693-x. PMID 31004126
- [Background] Xuan W, Agrawal T, Huang L, Gupta GK, Hamblin MR. Low-level laser therapy for traumatic brain injury in mice increases brain derived neurotrophic factor (BDNF) and synaptogenesis. J Biophotonics. 2015 Jun;8(6):502-11. doi: 10.1002/jbio.201400069. Epub 2014 Sep 8. PMID 25196192
- [Background] Xuan W, Vatansever F, Huang L, Hamblin MR. Transcranial low-level laser therapy enhances learning, memory, and neuroprogenitor cells after traumatic brain injury in mice. J Biomed Opt. 2014;19(10):108003. doi: 10.1117/1.JBO.19.10.108003. PMID 25292167
- [Background] Tian F, Hase SN, Gonzalez-Lima F, Liu H. Transcranial laser stimulation improves human cerebral oxygenation. Lasers Surg Med. 2016 Apr;48(4):343-9. doi: 10.1002/lsm.22471. Epub 2016 Jan 12. PMID 26817446
- [Background] Tedford CE, DeLapp S, Jacques S, Anders J. Quantitative analysis of transcranial and intraparenchymal light penetration in human cadaver brain tissue. Lasers Surg Med. 2015 Apr;47(4):312-22. doi: 10.1002/lsm.22343. Epub 2015 Mar 13. PMID 25772014
- [Background] Saltmarche AE, Naeser MA, Ho KF, Hamblin MR, Lim L. Significant Improvement in Cognition in Mild to Moderately Severe Dementia Cases Treated with Transcranial Plus Intranasal Photobiomodulation: Case Series Report. Photomed Laser Surg. 2017 Aug;35(8):432-441. doi: 10.1089/pho.2016.4227. Epub 2017 Feb 10. PMID 28186867
- [Background] Naeser MA, Saltmarche A, Krengel MH, Hamblin MR, Knight JA. Improved cognitive function after transcranial, light-emitting diode treatments in chronic, traumatic brain injury: two case reports. Photomed Laser Surg. 2011 May;29(5):351-8. doi: 10.1089/pho.2010.2814. Epub 2010 Dec 23. PMID 21182447
- [Background] Morries LD, Cassano P, Henderson TA. Treatments for traumatic brain injury with emphasis on transcranial near-infrared laser phototherapy. Neuropsychiatr Dis Treat. 2015 Aug 20;11:2159-75. doi: 10.2147/NDT.S65809. eCollection 2015. PMID 26347062
- [Background] Mester E, Spiry T, Szende B, Tota JG. Effect of laser rays on wound healing. Am J Surg. 1971 Oct;122(4):532-5. doi: 10.1016/0002-9610(71)90482-x. No abstract available. PMID 5098661
- [Background] Khuman J, Zhang J, Park J, Carroll JD, Donahue C, Whalen MJ. Low-level laser light therapy improves cognitive deficits and inhibits microglial activation after controlled cortical impact in mice. J Neurotrauma. 2012 Jan 20;29(2):408-17. doi: 10.1089/neu.2010.1745. Epub 2011 Sep 21. PMID 21851183
- [Background] Johnstone DM, Moro C, Stone J, Benabid AL, Mitrofanis J. Turning On Lights to Stop Neurodegeneration: The Potential of Near Infrared Light Therapy in Alzheimer's and Parkinson's Disease. Front Neurosci. 2016 Jan 11;9:500. doi: 10.3389/fnins.2015.00500. eCollection 2015. PMID 26793049
- [Background] Grillo SL, Duggett NA, Ennaceur A, Chazot PL. Non-invasive infra-red therapy (1072 nm) reduces beta-amyloid protein levels in the brain of an Alzheimer's disease mouse model, TASTPM. J Photochem Photobiol B. 2013 Jun 5;123:13-22. doi: 10.1016/j.jphotobiol.2013.02.015. Epub 2013 Mar 22. PMID 23603448
- [Background] Ferraresi C, Parizotto NA, Pires de Sousa MV, Kaippert B, Huang YY, Koiso T, Bagnato VS, Hamblin MR. Light-emitting diode therapy in exercise-trained mice increases muscle performance, cytochrome c oxidase activity, ATP and cell proliferation [J. Biophotonics 8, No. 9, 740-754 (2015)]. J Biophotonics. 2016 Sep;9(9):976. doi: 10.1002/jbio.201680087. Epub 2016 Jul 7. PMID 27592534
- [Background] undefined
- [Background] Eells JT, Henry MM, Summerfelt P, Wong-Riley MT, Buchmann EV, Kane M, Whelan NT, Whelan HT. Therapeutic photobiomodulation for methanol-induced retinal toxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3439-44. doi: 10.1073/pnas.0534746100. Epub 2003 Mar 7. PMID 12626762
- [Background] de Freitas LF, Hamblin MR. Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron. 2016 May-Jun;22(3):7000417. doi: 10.1109/JSTQE.2016.2561201. PMID 28070154
- [Background] Blanco NJ, Saucedo CL, Gonzalez-Lima F. Transcranial infrared laser stimulation improves rule-based, but not information-integration, category learning in humans. Neurobiol Learn Mem. 2017 Mar;139:69-75. doi: 10.1016/j.nlm.2016.12.016. Epub 2016 Dec 27. PMID 28039085
- [Background] Ayuk SM, Houreld NN, Abrahamse H. Effect of 660 nm visible red light on cell proliferation and viability in diabetic models in vitro under stressed conditions. Lasers Med Sci. 2018 Jul;33(5):1085-1093. doi: 10.1007/s10103-017-2432-2. Epub 2018 Mar 8. PMID 29520687
- [Background] Ando T, Xuan W, Xu T, Dai T, Sharma SK, Kharkwal GB, Huang YY, Wu Q, Whalen MJ, Sato S, Obara M, Hamblin MR. Comparison of therapeutic effects between pulsed and continuous wave 810-nm wavelength laser irradiation for traumatic brain injury in mice. PLoS One. 2011;6(10):e26212. doi: 10.1371/journal.pone.0026212. Epub 2011 Oct 18. PMID 22028832